CLINICAL TRIAL: NCT00966719
Title: The Impact of a Breastfeeding Support Intervention on Breastfeeding Duration in Jaundiced Infants Admitted to a Tertiary Care Centre: a Randomized Controlled Trial.
Brief Title: Breastfeeding Support Intervention in Jaundiced Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Catherine Pound, Consulting Pediatrician; Clinical Investigator, CHEO Research Institute, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 09/23E
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Jaundice; Breastfeeding
Keywords: Jaundice; Breastfeeding; Infants
MeSH Terms: conditions — Jaundice; Breast Feeding

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactation Consultant (Active Comparator): In hospital meeting with lactation consultant
  1 to 3 follow up visits at weekly intervals with lactation consultant
  Interventions: Other: Lactation Consultant support
- current treatment for jaundice (No Intervention): Babies will receive current standard of care for jaundice (IV fluids and phototherapy)

INTERVENTIONS:
Other: Lactation Consultant support — Meeting with lactation consultant once while in hospital and up to 3 times after discharge, in addition to current standard of care for jaundice.
  Other Names: Breastfeeding support
  Arms: Lactation Consultant

SUMMARY:
Breastfeeding decreases the risk of many infantile infectious diseases and certain types of cancers in women. It strengthens the bond between mothers and babies and decreases the health care cost to society by making children healthier. Although it is controversial, breastfeeding has been reported to increase the risk of jaundice in the neonatal period. There is some evidence that mothers of hospitalized jaundiced infants discontinue breastfeeding early, as they feel responsible for the baby's condition.

The main objective of this study is to determine the effect of a breastfeeding intervention on breastfeeding duration in jaundiced infants. All eligible infants will be randomized to one of two groups (an intervention or a control group). Mothers of infants in the intervention group will meet with a lactation consultant during their hospital stay, and three times post hospital discharge. Lactation consultants are individuals who have received certification in breastfeeding support from an international board, ensuring safe and effective practice. Mothers of infants in the control group will receive the current standard of care, which is typically support from the nursing staff, who are often not trained in lactation support. Information will be collected on length of time that infants are fed only breast milk, future visits to health care providers, mothers' need for breastfeeding support post hospital discharge, mothers' perception of their physicians' attitudes towards breastfeeding, and mothers' experiences at the hospital, as well as feedback on the intervention. Phone follow-up will occur one week post hospital discharge, and when the child is 2, 3, 4 and 6 months old.

The results of this study will clarify the importance of offering sound breastfeeding advice to mothers of young infants hospitalized with jaundice and help determine whether there is a need for trained lactation specialists in children's hospitals. It will allow us to examine whether such an intervention can have a quantifiable impact on children's health in their first 6 months of life, as measured by physician encounters and hospitalizations. It will also allow collection of information on advice and support given to breastfeeding women by primary care physicians, potentially identifying needs for more rigorous breastfeeding training during medical training.

DETAILED DESCRIPTION:
1.1 Overview This study will assess the effectiveness of a breastfeeding support intervention for infants admitted to the hospital with jaundice. It will evaluate the effect of this intervention on duration of breastfeeding and health care utilization.

1.2 Study Objectives: Primary: To determine the effect of a breastfeeding support intervention on breastfeeding duration in breastfeeding infants admitted to the hospital with jaundice.

Secondary:

* To determine the rate of breastfeeding failure, defined as breastfeeding cessation before the infant turns 6 months, in mothers of jaundiced infants randomized to the control group, as compared to the rate of breastfeeding failure in the general population.
* To compare subsequent healthcare utilization between groups during their first six months of life, as determined by the number of re-hospitalizations for jaundice, hospitalizations for non-jaundice related causes, as well as physician encounters.
* To determine the number of mothers seeking breastfeeding help once discharged from the hospital and compare it between both groups.
* To determine the kind and perceived effectiveness of breastfeeding support and advice given by the infant's primary physician throughout the child's first six months of life.

2.1 Summary: Breastfeeding confers many advantages to infants, mothers, families, and society in general. There is strong evidence that human milk feeding decreases the incidence of many infectious diseases and enhances the immunologic status of the newborn. It has been associated with enhanced performance on neurocognitive development tests, and has also been shown to provide important health benefits to the mother, including a decrease in risk of breast and ovarian cancers. It should be strongly encouraged for the first six months of life, and then continued for up to 2 years and beyond, as recommended in the World Health Organization's Innocent Declaration.

Neonatal jaundice is the most common problem in full-term infants during the immediate post-natal period. There is controversy as to whether breastfeeding increases the incidence of jaundice in the first days of life. In a study conducted in Italy, neonatal jaundice was not associated with breastfeeding per se, but rather with increased weight loss after birth subsequent to fasting, which can be seen with inadequate lactation.

When an infant is hospitalized, previously established patterns of breastfeeding are difficult to maintain. There is evidence to suggest that mothers of young infants admitted to hospital with hyperbilirubinemia commonly experience guilt as they feel breastfeeding caused the jaundice. Many of these women struggle with feelings of failure or inadequacy. A study recently conducted by the principal investigator of this current study (CP) suggested that infants admitted to the hospital with hyperbilirubinemia may have a higher rate of breastfeeding discontinuation than babies in the general population.

Previous studies have shown that breastfeeding support offered to various groups of mother-infant pairs significantly increased rates of breastfeeding at 2 to 6 months of age.

Given the clear health, social and economic advantages that breastfeeding confers to mothers, infants, and society in general, there is a need to assess the effectiveness of a breastfeeding support intervention for infants admitted to the hospital with jaundice.

2.2 Benefits of breastfeeding Breastfeeding is preferred for all infants, and exclusive breastfeeding of infants is recommended for the first 6 months after birth. Research has shown that human milk feeding decreases the incidence of multiple illnesses including bacterial meningitis, bacteremia, diarrhea, respiratory tract infection, otitis media, and urinary tract infections. A recent study conducted in Spain showed that exclusive breastfeeding lowered the risk of hospitalization as a result of infectious diseases during the first year of life. In that study, each additional month of exclusive breastfeeding would have avoided 30% of hospital admissions. A meta-analysis of 33 studies examining healthy infants in developed nations showed similar results, with formula-fed infants experiencing a tripling in severe respiratory illnesses compared with those who were exclusively breastfed for 4 months. Based on these results, breastfeeding promotion can lead to important economical gains from a societal perspective.

According to the most recent Ottawa Public Health Survey, breastfeeding rates in the general population are as follows: 91% of women initiate breastfeeding, with 56% practicing exclusive breastfeeding (no fluids other than breast milk). At 3 months, 71% of women continue to breastfeed, with 50% doing exclusive breastfeeding. This number drops to 60% for any breastfeeding at 6 months, with 39% of women exclusively breastfeeding.

2.3 Breastfeeding in hospitalized children Published reports have shown that previously established patterns of breastfeeding are hard to maintain once an infant is hospitalized. Moreover, as mentioned, evidence suggests that mothers of infants admitted to the hospital with jaundice experience guilt, as well feelings of failure and inadequacy as they often feel responsible for the child's admission to hospital. Maternal confidence has been shown to be a strong predictor of breastfeeding duration, with lack of confidence in breastfeeding skills leading to a higher likelihood of weaning in the first six weeks post-partum. There is only one study in the literature examining the rates of breastfeeding in the jaundiced population, which was done by the PI of this current study. Surveys were sent to all mothers of eligible infants admitted with jaundice to the Children's Hospital of Eastern Ontario (CHEO) over a 2.5 year period. One hundred and twenty-eight (64%) out of the 200 eligible mothers returned a completed survey. Of those, 92% had a post-secondary education. Information was collected, retrospectively, on length of breastfeeding after discharge from the hospital. Length of breastfeeding for hospitalized infants was compared to that of the Ottawa population, as reported by the City of Ottawa Public Health survey in 2005. Although numbers were the same between the jaundiced group and the City of Ottawa group, it is likely that the high education level of the study participants falsely elevated the rate of breastfeeding in the jaundiced infants. As mentioned, 92% of study participants had completed a post-secondary education, as compared to 53% of women involved in the population-based survey. Given that previous reports have shown that women with lower levels of education are more likely to discontinue breastfeeding early, it is reasonable to postulate that for comparable levels of education, mothers of infants admitted to the hospital with jaundice discontinue breastfeeding earlier than women in the general population.

2.4 Breastfeeding support interventions There are very few studies quantifying the effects of breastfeeding promotion interventions. A recent Cochrane review found that both professional and lay support were effective in prolonging breastfeeding. More specifically, this review found that professional support had more of an impact than lay support on both partial and exclusive breastfeeding and lay support affected exclusive breastfeeding. A review of four randomized controlled trials combining breastfeeding support with educational programs in developed countries found that combined education and support strategies increased short-term breastfeeding rates by 36%. Short-term breastfeeding in these studies was described as anywhere between 2 to 6 months. The education interventions were primarily conducted by lactation specialists or nurses as antepartum sessions, while the support interventions varied between telephone or in-person conversations, hospital or home visits by lactation consultants, nurses or peer counselors, and combined prearranged appointments and unscheduled visits or telephone calls for problems. Breastfeeding education and support had the biggest effect on initiation and maintenance of breastfeeding. Many of the studies however lacked scientific rigor. Most studies did not make a difference between exclusive and partial breastfeeding. Details regarding description and length of interventions as well as training of the individual delivering the educational session were often lacking.

A recent randomized controlled trial evaluating the effectiveness of a breastfeeding promotion intervention in the Republic of Belarus19 found an absolute increase of almost 37% in the prevalence of exclusive breastfeeding at 3 months in the intervention group. The chief obstetrician from each intervention maternity hospital, and the chief pediatrician from each intervention polyclinic, received the same 18-hour courses emphasizing methods to maintain lactation, promote exclusive and prolonged breastfeeding, and resolve common problems. All midwives, nurses and physicians providing care to study mothers and infants, as well as all pediatricians and nurses working in the polyclinics were trained over a period of 12 to 16 months. Such a program offered the advantage of providing reliable and consistent support, with the goal of being widely available. This study was published after the Cochrane review and thus is not included in the review.

Although no study published to date has determined which aspect of a breastfeeding support intervention yields positive results, it is likely to result from a combination of factors. Breastfeeding support results in increased confidence, and maternal confidence is known to be a strong predictor of breastfeeding outcome, with lack of confidence in breastfeeding skills leading to a higher likelihood of weaning in the first six weeks post-partum.

2.5 Availability of breastfeeding support In the recent CHEO study, 57% of the participating mothers needed to seek breastfeeding support after discharge from the hospital, suggesting they did not receive adequate help while hospitalized. Half of these women received help from private lactation consultants. These lactation consultants have variable training and may or may not hold recognized certifications or credentials. Their fees also vary from 10$ to 90$ an hour, and therefore may not be a suitable alternative for families with financial difficulties. This indicates the need for a standardized breastfeeding support intervention that will be accessible to all.

2.6 Breastfeeding and health care professionals Many studies have shown that physicians and physicians in training lack the necessary skills to offer proper guidance to lactating mothers. Freed et al surveyed pediatric residents and practitioners about breastfeeding knowledge and found that both groups had considerable knowledge deficits, and were ill-prepared for counseling mothers with lactation difficulties. Many residents surveyed in a study performed by Hillenbrand et al believed that early supplementation was not a cause of breast-feeding failure, although previous studies have clearly demonstrated this relationship. In the Ottawa study, only 3.9% of women reported receiving breastfeeding help from the treating physician while admitted to the hospital, suggesting the possibility that physicians do not have adequate knowledge to assess proper breastfeeding methods and counsel appropriately.

In summary, there is a need for this comprehensive study examining the impact of a breastfeeding support intervention for mothers of infants admitted to the hospital with jaundice. This study will clarify the rates of early breastfeeding discontinuation in the jaundiced population and help determine whether physicians in the Ottawa population have knowledge deficits when it comes to breastfeeding, as there may be a role for incorporating teaching of breastfeeding skills to physicians and physicians in training.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants admitted during the study period with hyperbilirubinemia, breastfeeding at the time of admission (any amount of breastfeeding)
* Mothers of infants < 1 month of age at the time of admission

Exclusion Criteria:

* Mothers of infants admitted with hyperbilirubinemia who are exclusively formula-fed
* Mothers of infants with hyperbilirubinemia of the predominantly conjugated type as this is a different disease, not associated with breastfeeding difficulties
* Mothers of infants with anatomical abnormalities, such as cleft lip or palate, as this would interfere with breastfeeding and require more intensive intervention.
* Mothers of neurologically impaired infants as breastfeeding may be more difficult in this population
* Mother of infants who were admitted to the Neonatal Intensive Care Unit (NICU) after birth and never went home as they are likely to have other comorbidities affecting feeding.
* Mothers of infants feeding via naso-gastric, naso-jejunal, or gastric tube
* Mothers of infants > 1 month of age
* Mothers who have had breast surgery in the past
* Foster mothers or adoptive mothers
* Mothers who do not understand English or French
* Mothers of infants that are the result of multiple birth (eg twins)

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2009-10; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Pound, MD, Principal Investigator — Children's Hospital of Eastern Ontario and Research Institute
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Gartner LM, Morton J, Lawrence RA, Naylor AJ, O'Hare D, Schanler RJ, Eidelman AI; American Academy of Pediatrics Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2005 Feb;115(2):496-506. doi: 10.1542/peds.2004-2491. PMID 15687461
- [Background] Heinig MJ. Host defense benefits of breastfeeding for the infant. Effect of breastfeeding duration and exclusivity. Pediatr Clin North Am. 2001 Feb;48(1):105-23, ix. doi: 10.1016/s0031-3955(05)70288-1. PMID 11236719
- [Background] Horwood LJ, Fergusson DM. Breastfeeding and later cognitive and academic outcomes. Pediatrics. 1998 Jan;101(1):E9. doi: 10.1542/peds.101.1.e9. PMID 9417173
- [Background] Anderson JW, Johnstone BM, Remley DT. Breast-feeding and cognitive development: a meta-analysis. Am J Clin Nutr. 1999 Oct;70(4):525-35. doi: 10.1093/ajcn/70.4.525. PMID 10500022
- [Background] Newcomb PA, Storer BE, Longnecker MP, Mittendorf R, Greenberg ER, Clapp RW, Burke KP, Willett WC, MacMahon B. Lactation and a reduced risk of premenopausal breast cancer. N Engl J Med. 1994 Jan 13;330(2):81-7. doi: 10.1056/NEJM199401133300201. PMID 8259187
- [Background] Collaborative Group on Hormonal Factors in Breast Cancer. Breast cancer and breastfeeding: collaborative reanalysis of individual data from 47 epidemiological studies in 30 countries, including 50302 women with breast cancer and 96973 women without the disease. Lancet. 2002 Jul 20;360(9328):187-95. doi: 10.1016/S0140-6736(02)09454-0. PMID 12133652
- [Background] Rosenblatt KA, Thomas DB. Lactation and the risk of epithelial ovarian cancer. The WHO Collaborative Study of Neoplasia and Steroid Contraceptives. Int J Epidemiol. 1993 Apr;22(2):192-7. doi: 10.1093/ije/22.2.192. PMID 8505173
- [Background] UNICEF-WHO. Innocenti Declaration. On the Protection, Promotion and Support of Breast-feeding. New York, NY:UNICEF;1990.
- [Background] Bertini G, Dani C, Tronchin M, Rubaltelli FF. Is breastfeeding really favoring early neonatal jaundice? Pediatrics. 2001 Mar;107(3):E41. doi: 10.1542/peds.107.3.e41. PMID 11230622
- [Background] Maisels MJ, Gifford K. Neonatal jaundice in full-term infants. Role of breast-feeding and other causes. Am J Dis Child. 1983 Jun;137(6):561-2. doi: 10.1001/archpedi.1983.02140320037007. PMID 6846290
- [Background] Schneider AP 2nd. Breast milk jaundice in the newborn. A real entity. JAMA. 1986 Jun 20;255(23):3270-4. PMID 3712679
- [Background] Rubaltelli FF. Unconjugated and conjugated bilirubin pigments during perinatal development. IV. The influence of breast-feeding on neonatal hyperbilirubinemia. Biol Neonate. 1993;64(2-3):104-9. doi: 10.1159/000243979. PMID 8260541
- [Background] Nielsen HE, Haase P, Blaabjerg J, Stryhn H, Hilden J. Risk factors and sib correlation in physiological neonatal jaundice. Acta Paediatr Scand. 1987 May;76(3):504-11. doi: 10.1111/j.1651-2227.1987.tb10507.x. PMID 3604669
- [Background] Willis SK, Hannon PR, Scrimshaw SC. The impact of the maternal experience with a jaundiced newborn on the breastfeeding relationship. J Fam Pract. 2002 May;51(5):465. PMID 12019058
- [Background] Pound CM, Gaboury I. The impact of jaundice in newborn infants on the length of breastfeeding. Paediatr Child Health. 2009 Sep;14(7):445-9. PMID 20808472
- [Background] Guise JM, Palda V, Westhoff C, Chan BK, Helfand M, Lieu TA; U.S. Preventive Services Task Force. The effectiveness of primary care-based interventions to promote breastfeeding: systematic evidence review and meta-analysis for the US Preventive Services Task Force. Ann Fam Med. 2003 Jul-Aug;1(2):70-8. doi: 10.1370/afm.56. PMID 15040435
- [Background] Kramer MS, Chalmers B, Hodnett ED, Sevkovskaya Z, Dzikovich I, Shapiro S, Collet JP, Vanilovich I, Mezen I, Ducruet T, Shishko G, Zubovich V, Mknuik D, Gluchanina E, Dombrovskiy V, Ustinovitch A, Kot T, Bogdanovich N, Ovchinikova L, Helsing E; PROBIT Study Group (Promotion of Breastfeeding Intervention Trial). Promotion of Breastfeeding Intervention Trial (PROBIT): a randomized trial in the Republic of Belarus. JAMA. 2001 Jan 24-31;285(4):413-20. doi: 10.1001/jama.285.4.413. PMID 11242425
- [Background] Canadian Paediatric Society, Dietitians of Canada and Health Canada. Nutrition for Healthy Term Infants. 1998. Ottawa: Minister of Public Works and Government Services, 1998
- [Background] Health Canada. Exclusive Breastfeeding Duration: 2004 Health Canada Recommendation. Ottawa, 2004. www.hc-sc.gc.ca/hpfb-dgpsa/onpp-bppn/exclusive_breastfeeding_duration_e.html
- [Background] World Health Organization. Global Strategy for Infant and Young Child Feeding, The Optimal Duration of Exclusive Breastfeeding. Geneva, 2001. www.who.int/gb/ebwha/pdf_files/WHA54/ea54id4.pdf
- [Background] Cochi SL, Fleming DW, Hightower AW, Limpakarnjanarat K, Facklam RR, Smith JD, Sikes RK, Broome CV. Primary invasive Haemophilus influenzae type b disease: a population-based assessment of risk factors. J Pediatr. 1986 Jun;108(6):887-96. doi: 10.1016/s0022-3476(86)80922-2. PMID 3712153
- [Background] Istre GR, Conner JS, Broome CV, Hightower A, Hopkins RS. Risk factors for primary invasive Haemophilus influenzae disease: increased risk from day care attendance and school-aged household members. J Pediatr. 1985 Feb;106(2):190-5. doi: 10.1016/s0022-3476(85)80285-7. PMID 3871478
- [Background] Takala AK, Eskola J, Palmgren J, Ronnberg PR, Kela E, Rekola P, Makela PH. Risk factors of invasive Haemophilus influenzae type b disease among children in Finland. J Pediatr. 1989 Nov;115(5 Pt 1):694-701. doi: 10.1016/s0022-3476(89)80644-4. PMID 2809900
- [Background] Dewey KG, Heinig MJ, Nommsen-Rivers LA. Differences in morbidity between breast-fed and formula-fed infants. J Pediatr. 1995 May;126(5 Pt 1):696-702. doi: 10.1016/s0022-3476(95)70395-0. PMID 7751991
- [Background] Howie PW, Forsyth JS, Ogston SA, Clark A, Florey CD. Protective effect of breast feeding against infection. BMJ. 1990 Jan 6;300(6716):11-6. doi: 10.1136/bmj.300.6716.11. PMID 2105113
- [Background] Popkin BM, Adair L, Akin JS, Black R, Briscoe J, Flieger W. Breast-feeding and diarrheal morbidity. Pediatrics. 1990 Dec;86(6):874-82. PMID 2251024
- [Background] Lopez-Alarcon M, Villalpando S, Fajardo A. Breast-feeding lowers the frequency and duration of acute respiratory infection and diarrhea in infants under six months of age. J Nutr. 1997 Mar;127(3):436-43. doi: 10.1093/jn/127.3.436. PMID 9082027
- [Background] Bachrach VR, Schwarz E, Bachrach LR. Breastfeeding and the risk of hospitalization for respiratory disease in infancy: a meta-analysis. Arch Pediatr Adolesc Med. 2003 Mar;157(3):237-43. doi: 10.1001/archpedi.157.3.237. PMID 12622672
- [Background] Oddy WH, Sly PD, de Klerk NH, Landau LI, Kendall GE, Holt PG, Stanley FJ. Breast feeding and respiratory morbidity in infancy: a birth cohort study. Arch Dis Child. 2003 Mar;88(3):224-8. doi: 10.1136/adc.88.3.224. PMID 12598384
- [Background] Duncan B, Ey J, Holberg CJ, Wright AL, Martinez FD, Taussig LM. Exclusive breast-feeding for at least 4 months protects against otitis media. Pediatrics. 1993 May;91(5):867-72. PMID 8474804
- [Background] Aniansson G, Alm B, Andersson B, Hakansson A, Larsson P, Nylen O, Peterson H, Rigner P, Svanborg M, Sabharwal H, et al. A prospective cohort study on breast-feeding and otitis media in Swedish infants. Pediatr Infect Dis J. 1994 Mar;13(3):183-8. doi: 10.1097/00006454-199403000-00003. PMID 8177624
- [Background] Marild S, Hansson S, Jodal U, Oden A, Svedberg K. Protective effect of breastfeeding against urinary tract infection. Acta Paediatr. 2004 Feb;93(2):164-8. doi: 10.1080/08035250310007402. PMID 15046267
- [Background] Pisacane A, Graziano L, Zona G. Breastfeeding and urinary tract infection. Lancet. 1990 Jul 7;336(8706):50. doi: 10.1016/0140-6736(90)91559-s. No abstract available. PMID 1973227
- [Background] Paricio Talayero JM, Lizan-Garcia M, Otero Puime A, Benlloch Muncharaz MJ, Beseler Soto B, Sanchez-Palomares M, Santos Serrano L, Rivera LL. Full breastfeeding and hospitalization as a result of infections in the first year of life. Pediatrics. 2006 Jul;118(1):e92-9. doi: 10.1542/peds.2005-1629. PMID 16818542
- [Background] City of Ottawa, Ottawa Public Health. Infant Care Survey 2005
- [Background] Britton C, McCormick FM, Renfrew MJ, Wade A, King SE. Support for breastfeeding mothers. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD001141. doi: 10.1002/14651858.CD001141.pub3. PMID 17253455
- [Background] Freed GL, Clark SJ, Sorenson J, Lohr JA, Cefalo R, Curtis P. National assessment of physicians' breast-feeding knowledge, attitudes, training, and experience. JAMA. 1995 Feb 8;273(6):472-6. doi: 10.1001/jama.1995.03520300046035. PMID 7837365
- [Background] Williams EL, Hammer LD. Breastfeeding attitudes and knowledge of pediatricians-in-training. Am J Prev Med. 1995 Jan-Feb;11(1):26-33. PMID 7748583
- [Background] Hillenbrand KM, Larsen PG. Effect of an educational intervention about breastfeeding on the knowledge, confidence, and behaviors of pediatric resident physicians. Pediatrics. 2002 Nov;110(5):e59. doi: 10.1542/peds.110.5.e59. PMID 12415065
- [Background] Olson CM, Psiaki DL. Imparting information on breastfeeding to medical students. J Med Educ. 1978 Oct;53(10):845-7. doi: 10.1097/00001888-197810000-00010. No abstract available. PMID 712774
- [Background] Wright A, Rice S, Wells S. Changing hospital practices to increase the duration of breastfeeding. Pediatrics. 1996 May;97(5):669-75. PMID 8628605
- [Background] Sadeharju K, Knip M, Virtanen SM, Savilahti E, Tauriainen S, Koskela P, Akerblom HK, Hyoty H; Finnish TRIGR Study Group. Maternal antibodies in breast milk protect the child from enterovirus infections. Pediatrics. 2007 May;119(5):941-6. doi: 10.1542/peds.2006-0780. PMID 17473095
- [Background] Wright AL, Holberg CJ, Martinez FD, Morgan WJ, Taussig LM. Breast feeding and lower respiratory tract illness in the first year of life. Group Health Medical Associates. BMJ. 1989 Oct 14;299(6705):946-9. doi: 10.1136/bmj.299.6705.946. PMID 2508946
- [Background] von Kries R, Koletzko B, Sauerwald T, von Mutius E, Barnert D, Grunert V, von Voss H. Breast feeding and obesity: cross sectional study. BMJ. 1999 Jul 17;319(7203):147-50. doi: 10.1136/bmj.319.7203.147. PMID 10406746
- [Derived] Pound CM, Moreau K, Rohde K, Barrowman N, Aglipay M, Farion KJ, Plint AC. Lactation support and breastfeeding duration in jaundiced infants: a randomized controlled trial. PLoS One. 2015 Mar 6;10(3):e0119624. doi: 10.1371/journal.pone.0119624. eCollection 2015. PMID 25747308

RESULTS

PARTICIPANT FLOW:
Groups:
- Lactation Consultant: In hospital meeting with lactation consultant
  1 to 3 follow up visits at weekly intervals with lactation consultant
  Lactation Consultant support: Meeting with lactation consultant once while in hospital and up to 3 times after discharge, in addition to current standard of care for jaundice.
Period: Overall Study
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Started | 50 | 49
Completed | 44 | 38
Not Completed | 6 | 11
Not completed — Lost to Follow-up | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactation Consultant | Current Treatment for Jaundice | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Customized [Number; unit: participants]
  15-20 years | 2 | 0 | 2
  21-25 years | 6 | 9 | 15
  26-30 years | 11 | 13 | 24
  31-35 years | 23 | 18 | 41
  36-40 years | 6 | 7 | 13
  >40 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 99
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
language [Number; unit: participants]
  English | 50 | 43 | 93
  French | 0 | 6 | 49
highest level of education completed [Count of Participants; unit: Participants]
  Completed high school | 4 | 4 | 8
  Vocational / technical training (post high school) | 13 | 13 | 26
  Some university training | 5 | 4 | 9
  Completed university | 28 | 28 | 56
combined household income [Count of Participants; unit: Participants]
  Under $30,000 | 4 | 7 | 11
  $30,000 - $69,000 | 8 | 9 | 17
  $70,000 - $100,000 | 10 | 12 | 22
  Above $100,000 | 21 | 18 | 39
  Declined to answer | 6 | 2 | 8
mother smokes at home [Count of Participants; unit: Participants] | 1 | 0 | 1
marital status [Count of Participants; unit: Participants]
  marries / common-law | 45 | 47 | 92
  single | 5 | 1 | 6
  unknown | 0 | 1 | 1
number of prior children [Count of Participants; unit: Participants]
  none | 22 | 31 | 53
  1 | 22 | 14 | 36
  >1 | 6 | 8 | 14
number of prior breastfed children [Count of Participants; unit: Participants]
  0 | 24 | 31 | 55
  1 | 23 | 15 | 38
  >1 | 3 | 3 | 6
received breastfeeding support with prior infants [Count of Participants; unit: Participants] | 14 | 15 | 29
infant received formula prior to hospitalization [Count of Participants; unit: Participants] | 27 | 22 | 49
received medical care from: [Number; unit: participants]
  obstetrician | 32 | 29 | 61
  family physician | 29 | 21 | 50
  midwife | 8 | 15 | 23
  no prenatal care | 3 | 0 | 3
attended prenatal classes [Count of Participants; unit: Participants] | 17 | 21 | 38
planning to return to work before child is 1 year of age [Count of Participants; unit: Participants] | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Exclusively Breastfeeding at 3 Months, or 3 Months Corrected if the Infant Was Born Prematurely
Description: Exclusive breastfeeding was defined as no milk intake other than breast milk
Time Frame: 3 months
Population: 50 randomized to intervention; by 3 months 5 lost to follow up (45). By 6 months, 1 more patient lost to follow up (44), as reported in Participant Flow Module
  49 randomized to control group; by 3 months 8 lost to follow up (41). By 6 months, 3 more patients lost to follow up (38), as reported in Participant Flow Module
Measure: Count of Participants; unit: Participants
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Number analyzed (Participants) | 45 | 41
Participants | 22 | 24
Statistical Analysis 1: Comparison: Lactation Consultant vs Current Treatment for Jaundice; Test type: Other; p = 0.40, Fisher Exact; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.56 to 1.24]

2. Secondary Outcome: Number of Participants Exclusively Breastfeeding at 6 Months, or 6 Months Corrected if the Infant Was Born Prematurely
Description: Exclusive breastfeeding was defined as no milk intake other than breast milk
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Number analyzed (Participants) | 44 | 38
Participants | 8 | 6
Statistical Analysis 1: Comparison: Lactation Consultant vs Current Treatment for Jaundice; Test type: Other; p = 1, Fisher Exact; Risk Ratio (RR) = 1.15, 95% CI 2-sided [0.44 to 3.02]

3. Secondary Outcome: Number of Participants Partially Breastfeeding at 3 Months, or 3 Months Corrected if the Infant Was Born Prematurely
Description: Partial breastfeeding was defined as any feeding of breast milk
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Number analyzed (Participants) | 45 | 41
Participants | 43 | 39
Statistical Analysis 1: Comparison: Lactation Consultant vs Current Treatment for Jaundice; Test type: Other; p = 1, Fisher Exact; Risk Ratio (RR) = 1, 95% CI 2-sided [0.91 to 1.10]

4. Secondary Outcome: Number of Participants Partially Breastfeeding at 6 Months, or 6 Months Corrected if the Infant Was Born Prematurely
Description: Partial breastfeeding was defined as any amount of feeding breast milk
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Number analyzed (Participants) | 44 | 38
Participants | 37 | 31
Statistical Analysis 1: Comparison: Lactation Consultant vs Current Treatment for Jaundice; Test type: Other; p = 0.78, Fisher Exact; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.85 to 1.26]

5. Secondary Outcome: Number of Participants With an Infant Re-hospitalized for Jaundice
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Number analyzed (Participants) | 50 | 49
Participants | 3 | 1
Statistical Analysis 1: Comparison: Lactation Consultant vs Current Treatment for Jaundice; Test type: Other; p = 0.32, Fisher Exact; Risk Ratio (RR) = 2.94, 95% CI 2-sided [0.32 to 27.30]

6. Secondary Outcome: Number of Participants With an Infant Re-hospitalized for Non-jaundice Related Causes in the First Six Months of Life
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Number analyzed (Participants) | 50 | 49
Participants | 2 | 3
Statistical Analysis 1: Comparison: Lactation Consultant vs Current Treatment for Jaundice; Test type: Other; p = 0.09, Fisher Exact; Risk Ratio (RR) = 1.50, 95% CI 2-sided [0.95 to 2.38]

7. Secondary Outcome: Number of Physician Encounters in First 6 Months of Life
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: physician encounters
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Number analyzed (Participants) | 50 | 49
physician encounters | 9.2 [6 to 12] | 9.9 [6.3 to 12]
Statistical Analysis 1: Comparison: Lactation Consultant vs Current Treatment for Jaundice; Test type: Other; p = 0.77, Fisher Exact; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.83 to 1.27]

8. Secondary Outcome: Number of Mothers Seeking Breastfeeding Help
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Number analyzed (Participants) | 44 | 38
Participants | 11 | 7
Statistical Analysis 1: Comparison: Lactation Consultant vs Current Treatment for Jaundice; Test type: Other; p = 0.6, Fisher Exact; Risk Ratio (RR) = 1.36, 95% CI 2-sided [0.58 to 3.15]

ADVERSE EVENTS:
Arm/Group | Lactation Consultant | Current Treatment for Jaundice
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49

LIMITATIONS AND CAVEATS:
Difficult recruitment Large CI around our risk ratio (0.56 to 1.24) for primary outcome women with a strong desire to breastfeed more likely to enrol (breastfeeding proportions in control much higher than in general population).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes